CLINICAL TRIAL: NCT04779268
Title: Large Scale ICU Data Sharing for 1000 Critically Ill Patients With Severe Respiratory Distress Syndrome Coronavirus in Three Distinct Isolation Centers
Brief Title: Large Scale ICU Data Sharing for 1000 Critically Ill Patients With Severe Acute Respiratory Distress Syndrome Coronavirus (SARS.COV19) in Three Distinct Isolation Centers
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, Lecturer of anesthesia and ICU, Minia University
Other Study IDs: 181/2-2021
Record Dates: First submitted 2021-02-23; First posted 2021-03-03 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Median Nerve Entrapement
Keywords: neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cohort study of patients with severe respiratory distress syndrome coronavirus2 in three different isolation hospitals recording data about outcome.

ELIGIBILITY:
Inclusion Criteria:

* All COVID positive candidates

Exclusion Criteria:

* patient refusal

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID positive patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
follow up | 3 months
  mortality, length of ICU stay, ( days)

SECONDARY OUTCOMES:
prediction | 3 months
  prediction of mortality and morbidity

CONTACTS AND LOCATIONS:
Locations (1):
- Mina Raouf, Minya, Minya Governorate, Egypt